CLINICAL TRIAL: NCT04006223
Title: The Diagnostic Value of Hybrid PET/MR for Systemic Amyloidosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoli Lan, Director of the Department of nuclear medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: XLan-S895
Record Dates: First submitted 2019-06-30; First posted 2019-07-05 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Systemic Amyloidosis; PET/MR
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 11C-PIB or 18F-florbetapir PET/MR: Patients suspected of or diagnosed with systemic amyloidosis will be scanned by 11C-PIB or 18F-florbetapir PET/MR twice. One is before biopsy and treatment, and the other is after at least half a year of treatment.
  Interventions: Diagnostic Test: 11C-PIB or 18F-florbetapir PET/MR before biopsy and treatment; Diagnostic Test: 11C-PIB or 18F-florbetapir PET/MR after treatment

INTERVENTIONS:
Diagnostic Test: 11C-PIB or 18F-florbetapir PET/MR before biopsy and treatment — 10-20 mCi 11C-PIB or 5-10 mCi 18F-florbetapir will be injected intravenously prior to imaging.
Diagnostic Test: 11C-PIB or 18F-florbetapir PET/MR after treatment — 10-20 mCi 11C-PIB or 5-10 mCi 18F-florbetapir will be injected intravenously prior to imaging.

SUMMARY:
Systemic amyloidosis is a multi-system disease caused by extracellular deposition of insoluble amyloid fibrils in various tissues and organs, leading to progressive organ dysfunction. The clinical manifestations of different types of amyloidosis are complex and diverse, and the prognosis is very poor. Early detection and classification of amyloid deposition is becoming increasingly important. However, conventional imaging techniques including ultrasound and magnetic resonance are not sensitive or specific. Endocardial biopsy is the gold standard for the diagnosis of cardiac amyloidosis, but it is an invasive procedure with a clinical complication rate of 6%.

Positron emission tomography (PET) provides a valuable tool for diagnosing systemic amyloidosis. Recently, amyloid PET imaging agents (11C-PIB or 18F-florbetapir) have been shown to be effective as novel positron tracers to detect potential amyloid deposition in some small sample studies. The investigators will use the most advanced imaging equipment, integrated PET/MR with amyloid PET imaging agents(11C-PIB or 18F-florbetapir) to image patients suspected or confirmed systemic amyloidosis, the aim is to explore the value of hybrid PET/MR for systemic amyloidosis.

DETAILED DESCRIPTION:
Systemic amyloidosis is a multi-system disease caused by extracellular deposition of insoluble amyloid fibrils in various tissues and organs, leading to progressive organ dysfunction. The clinical manifestations of different types of amyloidosis are complex and diverse, and the prognosis is very poor. Early detection and classification of amyloid deposition is becoming increasingly important. However, conventional imaging techniques including ultrasound and magnetic resonance are not sensitive or specific. Endocardial biopsy is the gold standard for the diagnosis of cardiac amyloidosis, but it is an invasive procedure with a clinical complication rate of 6%.

Positron emission tomography (PET) provides a valuable tool for diagnosing systemic amyloidosis. Recently, amyloid PET imaging agents (11C-PIB or 18F-florbetapir) have been shown to be effective as novel positron tracers to detect potential amyloid deposition in multiple organs in some small sample studies. The investigators will use the most advanced imaging equipment, integrated PET/MR with amyloid PET imaging agents(11C-PIB or 18F-florbetapir) to image patients suspected or confirmed systemic amyloidosis, the aim is to explore the value of hybrid PET/MR for systemic amyloidosis.

For patients suspected of or diagnosed with systemic amyloidosis, the investigators aim to evaluate the roles of hybrid PET/MR in differential diagnosis, detecting the deposition of amyloid in various tissues and organs of the body, guiding biopsy, and determining treatment plan prior to treatment; for the patients with a history of systemic amyloidosis, the aim is to evaluate the value of hybrid PET/MR for treatment response assessment.

ELIGIBILITY:
Inclusion Criteria:

Patient with Monoclonal Ganunopathy, adds one of the following criteria:

* Histologically confirmed Amyloidosis of any organ.
* Average left ventricular thickness of the echocardiogram is more than 11 mm without uncontrolled high blood pressure.
* 12-lead ECG shows unexplained low voltage <0.5 mV.

Exclusion Criteria:

* Patient can not lie flat
* NYHA Level 4 Heart Failure
* Patient is pregnant or nursing
* Patient is allergic to amyloid PET imaging agents
* Patient with acute systemic diseases and electrolyte disorders
* Patient with severe claustrophobia or unstable vital sigh
* Other serious comorbidities evaluated by primary investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Central China
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity per patient analysis | up to 2 years
  For patient without any treatment, detection and initial diagnosis, results of 11C-PiB or 18F-florbetapir PET/MR will be compared to histopathological, clinical, laboratory, radiological evidence and follow-up result.

SECONDARY OUTCOMES:
Sensitivity and specificity per organ analysis | up to 2 years
  For patient without any treatment, detection and initial diagnosis, results of 11C-PiB or 18F-florbetapir PET/MR will be compared to histopathological, clinical, laboratory, radiological evidence and follow-up result.
Change after treatment | up to 2 years
  For patient after treatment, change of PET/MR scan and clinical/radiological/histopathological indices.
Correlation with severity | up to 2 years
  Correlation of 11C-PiB or 18F-florbetapir uptake with clinical/radiological/histopathological indices of amyloidosis severity.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, MD, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- China, Hubei Province, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided